CLINICAL TRIAL: NCT00121706
Title: Fast Food Feeding in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: P30DK040561 (NIH)
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2006-02-06 (Estimated); Status verified 2006-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Condition A (see detailed summary)
Behavioral: Condition B (see detailed summary)
Behavioral: Condition C (see detailed summary)

SUMMARY:
The primary aim of the proposed pilot study is to assess the effects of fast food meals, varying in serving size and rate of delivery, on energy (calorie) intake in adolescents.

DETAILED DESCRIPTION:
Using a three-period crossover design, the investigators will evaluate three acute feeding conditions.

* Under Condition A, the total amount of food in a large fast food meal will be delivered on a single tray at Time 0 (start of meal).
* Under Condition B, the same fast food meal will be equally divided among 4 separate portions, with all portions delivered at Time 0.
* Under Condition C, the meal again will be equally divided among 4 separate portions, but the portions will be delivered at 15-minute time intervals (Time 0, 15 minutes, 30 minutes, 45 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between the 85th and 98th percentiles for sex and age
* Consumption of fast food at least one time per week
* Willingness to eat the foods specified in the research methods
* Parent/guardian willing and able to cooperate
* Access to a working telephone

Exclusion Criteria:

* Major medical illness (eg, diabetes; heart, renal, or liver disease; cancer; endocrinopathy)
* Taking any prescription medication that may affect food intake
* Current smoking (i.e., any tobacco in the last month)
* Previous diagnosis of an eating disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18
Dates: Start 2005-07; Study Completion 2005-09

PRIMARY OUTCOMES:
Energy (calorie) intake during fast food feedings, assessed by direct observation

SECONDARY OUTCOMES:
Energy (calorie) intake during the day of the visit and the day after the visit, assessed by multiple-pass dietary recall interview methodology

CONTACTS AND LOCATIONS:
Overall Officials: Cara B Ebbeling, PhD, Principal Investigator — Boston Children's Hospital; David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ebbeling CB, Sinclair KB, Pereira MA, Garcia-Lago E, Feldman HA, Ludwig DS. Compensation for energy intake from fast food among overweight and lean adolescents. JAMA. 2004 Jun 16;291(23):2828-33. doi: 10.1001/jama.291.23.2828. PMID 15199032